CLINICAL TRIAL: NCT02073318
Title: Effects of Task-oriented Balance Training in Institutionalized Older Adults With Dementia
Brief Title: Effects of Balance Training in Older Adults With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201011010RB
Record Dates: First submitted 2011-01-20; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance training (Experimental)
  Interventions: Other: Task-oriented balance training
- Control (Active Comparator): Control group received 4 weeks upper extremities exercise in sitting position
  Interventions: Other: Upper extremities exercise

INTERVENTIONS:
Other: Task-oriented balance training — 4 weeks individualized task-oriented balance training, twice a week and 1 hour each session
  Arms: Balance training
Other: Upper extremities exercise — 4 weeks upper extremities exercise in sitting position, twice a week and 1 hour each session
  weeks
  Arms: Control

SUMMARY:
Purpose -To investigate whether older adults with dementia who have balance and gait problems can improve their balance and gait function after an individualized 4-week tasks-oriented balance training with sensory manipulation.

Hypothesis

-There is significant difference of Timed Up and Go Test, Berg Balance Scale, walking speed, 30-s chair-stand test, Chair sit-and-reach test and Barthel Index between dementia patients who received tasks-oriented balance training and those didn't receive after 4-weeks training and one month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides oral consent, and written consent obtains from next of kin
* Older than 65 years
* Diagnosis of dementia, based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) or The International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10)
* Can follow order to complete the screening test(Timed Up and Go test)
* Has balance and gait problems
* Can standing independently with/without assistive device or can standing with minimal assistance

Exclusion Criteria:

* Newly developed cardiopulmonary disease and other exercise contraindications
* Other neuromuscular or musculoskeletal disease that might affect the outcome(ex. Recent stroke, fracture or orthopedic surgery)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test | baseline, post-treatment, 1-month follow up
  Change from Baseline of Timed Up and Go test
Berg Balance Scale | baseline, post-treatment, 1-month follow up
  Change from Baseline of Berg Balance Scale
walking speed | baseline, post-treatment, 1-month follow up
  Change from Baseline of walking speed

SECONDARY OUTCOMES:
30-s chair-stand test | baseline, post-treatment, 1-month follow up
  Change from Baseline of 30-s chair-stand test
chair sit-and-reach test | baseline, post-treatment, 1-month follow up
  Change from Baseline of chair sit-and-reach test
Saint Louis University mental status examination | baseline, post-treatment, 1-month follow up
  Change from Baseline of Saint Louis University mental status examination
Barthel index | baseline, post-treatment, 1-month follow up
  Change from Baseline of Barthel index

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hsia Hu, Ph.D., Study Chair — School of Physical Therapy, National Taiwan University
Locations (1):
- The Catholic Foundation of Alzheimer's Disease and Related Dementia St. Joseph Home for Alzheimer's Disease and Related Dementia, Taipei, Taipei, Taiwan